CLINICAL TRIAL: NCT01693120
Title: Evaluation of Multielectrode Phased RF Technology in Persistent Atrial Fibrillation
Brief Title: Evaluation of the Phased Radio Frequency Ablation System
Acronym: VICTORY-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped solely based on lower than expected enrollment rate.
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICTORY AF
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Persistent Atrial Fibrillation
Keywords: ablation; atrial fibrillation; Radio frequency
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Treatment with Phased RF Ablation System
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ablation (Experimental): Phased RF ablation
  Interventions: Device: Medtronic Phased RF Ablation System

INTERVENTIONS:
Device: Medtronic Phased RF Ablation System — Phased RF ablation

SUMMARY:
VICTORY AF is an IDE, prospective global, multi-center, single arm, controlled, unblinded, investigational clinical study. The purpose of this clinical study is to evaluate the risk of procedure and/or device related strokes in subjects with persistent or long-standing persistent atrial fibrillation (AF) undergoing ablation with the Phased RF System.

ELIGIBILITY:
Inclusion Criteria:

* History of symptomatic persistent or long-standing persistent atrial fibrillation
* Failure of at least one anti-arrhythmic drug

Exclusion Criteria:

* Structural heart disease
* Prior ablation in left atrium for AF
* Known sensitivities (or allergy) to heparin, warfarin, contrast media
* Contraindicated for MRI
* Invasive cardiovascular procedure performed or planned within 3 month period of ablation procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-11; Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hummel, MD, Principal Investigator — Ohio State University
Locations (40):
- United States (31):
  - Phoenix Cardiovascular - Banner, Phoenix, Arizona
  - Hoag Hospital, Newport Beach, California
  - Medical Center of the Rockies, Fort Collins, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - St. Vincent's Ambulatory Care, Jacksonville, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Northwestern University, Chicago, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - DLP Marquette Physicians Practice, Marquette, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - HealthEast St Joseph's Hospital, Saint Paul, Minnesota
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Asheville Cardiology, Asheville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Doylestown Cardiology - VIAA, Doylestown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Baylor Research Institute - Dallas, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Baylor Research Institute - Plano, Plano, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Swedish Medical Center - Cherry Hill, Seattle, Washington
- Canada (3):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Hopital du Sacre Coeur de Montreal, Montreal, Quebec
- Debreceni Egyetem, Debrecen, Hungary
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
- United Kingdom (3):
  - Basildon and Thurrock University Hospitals, Basildon
  - Blackpool, Fylde and Wyre Hospitals, Blackpool
  - Newcastle Upon Tyne Hospitals, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 05 November 2013 and the first Phased RF procedure occurred on 17 December 2013. Enrollment into the VICTORY AF study was closed on 26 June 2016 prior to reaching the target sample size due to slower than expected enrollment rate.
Period: Enrollment
Arm/Group | Ablation
Started | 199 (70 subjects exited the study after consent, but prior to undergoing a study ablation procedure.)
Completed | 129 (129 of the 199 enrolled subjects underwent a Phased RF study procedure)
Not Completed | 70
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 10
Not completed — Protocol Violation | 46
Not completed — Physician Decision | 3
Not completed — Adverse Event | 1
Not completed — Study closed | 8
Not completed — Other | 1
Period: Phased RF Study Procedure and Follow-up
Arm/Group | Ablation
Started | 129
Completed | 112 (112 of the 129 subjects with a Phased RF procedure completed the 6-month follow-up visit)
Not Completed | 17
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 1
Not completed — Other reasons | 7

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is the number of subjects that had an ablation attempt with the Phased RF system.
Arm/Group | Ablation
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 123
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Canada | 10
  Netherlands | 13
  Hungary | 5
  United States | 94
  United Kingdom | 7
Atrial fibrillation type [Count of Participants; unit: Participants]
  persistent atrial fibrillation | 108
  long-term persistent atrial fibrillation | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedure and/or Device Related Stroke
Description: A stroke with with a symptom onset date within 30 days of an ablation procedure where at least one Phased RF ablation catheter was deployed into the left atrium considered related to the procedure and/or the investigational device by the independent clinical events committee
Time Frame: 30 days
Population: All subjects with a Phased RF ablation procedure who did not have a non-investigational catheter placed in the left atrium
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation
Number analyzed (Participants) | 127
Participants | 2
Statistical Analysis 1: Comparison: Ablation; The null hypothesis was that the procedure or device related stroke rate within 30-days of a Phased RF ablation procedure was 3.5% or greater. The alternative hypothesis was that this rate was less than 3.5%. A sample size of 300 subjects provided 90% power to test the null hypothesis assuming the true stroke rate was 1.0% with a one-sided type I error rate of 0.05; Test type: Superiority; p = 0.175, exact binomial test; rate = 1.6, 95% CI 1-sided [upper limit 4.9]

2. Secondary Outcome: 6-month Post-procedure Effectiveness
Description: For a participant, the 6-month effectiveness defined as meeting all of the following criteria: (1) acute procedural success, (2) greater than 90% reduction in atrial fibrillation/atrial flutter episodes lasting longer than 10 minutes as measured by 48-hour ambulatory ECG, (3) No amiodarone use for 90 days and no class I or class III antiarrhythmic drugs for at least 60 days prior to 6-month ambulatory ECG, and (4) free from direct current cardioversion for at least 60 days prior to the 6-month ambulatory ECG
Time Frame: 6 months
Population: Of the 129 subjects with an index Phased RF ablation procedure, 114 were evaluable for the 6-month efficacy objective. There were 15 subjects that were not included in the 6-month efficacy objective; 13 due to study exit prior to the 6-month visit and 2 due to no 6-month ambulatory ECG
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation
Number analyzed (Participants) | 114
Participants | 60
Statistical Analysis 1: Comparison: Ablation; Test type: Other — The goal of the analysis was to compute a two-sided 95% confidence interval around the 6-month effectiveness rate. There was no pre-specified hypothesis; rate = 52.6, 95% CI 2-sided [43.1 to 62.1]

3. Secondary Outcome: Number of Participants With Acute Procedural Success
Description: Acute procedural success defined as: (1) Only Phased RF ablation catheters used in the left atrium, (2) all targeted pulmonary veins isolated, (3) all complex fractionated atrial electrograms and high frequency intracardiac electrogram amplitudes were mapped and ablated, and (4) sinus rhythm was restored at the end of the ablation procedure (with or without cardioversion)
Time Frame: 30 minutes
Population: All subjects who underwent a Phased RF study procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation
Number analyzed (Participants) | 129
Participants | 117
Statistical Analysis 1: Comparison: Ablation; There was no prespecified hypothesis tested; Test type: Other — There was no prespecified hypothesis tested; rate = 90.7, 95% CI 2-sided [84.3 to 95.1]

4. Secondary Outcome: Number of Participants With Pulmonary Vein Stenosis
Description: Greater than 70 percent reduction in the luminal diameter in any one or more of the pulmonary veins following a Phased RF ablation procedure
Time Frame: 3 months
Population: Number of subjects selected for participation in the pulmonary vein assessment cohort with baseline and 3-month evaluable magnetic resonance imaging scans of the pulmonary veins
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation
Number analyzed (Participants) | 59
Participants | 0
Statistical Analysis 1: Comparison: Ablation; There was no pre-specified hypothesis to test; Test type: Other — There was no pre-specified hypothesis to test; rate = 0, 95% CI 2-sided [0 to 6.1]

ADVERSE EVENTS:
Time Frame: All adverse events were collected between subject consent and study completion (6-months post Phased RF study ablation procedure) or study exit
Arm/Group | Ablation
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 28/129
Other Adverse Events (participants affected / at risk) | 38/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation (N=129)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 5 (5)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation (N=129)
Visual impairment (Eye disorders) | 4 (4)
Chest discomfort (General disorders) | 4 (4)
Chest pain (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 5 (5)
Influenza (Infections and infestations) | 4 (4)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 5 (5)
Dizziness (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 10 (10)
Haematuria (Renal and urinary disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
The study stopped enrolling prematurely due to slow enrollment. Since the achieved sample size is 57% smaller than the planned sample size of 300 evaluable subjects, the study objectives could not be properly evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2014-11-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT01693120/Prot_000.pdf
  • Statistical Analysis Plan (2013-07-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT01693120/SAP_001.pdf